CLINICAL TRIAL: NCT01176864
Title: Prospective Trial Comparing Push-and-Pull Enteroscopy With the Single- and Double-Balloon Techniques in Patients With Obscure Small-Bowel Bleeding
Brief Title: Double- Versus Single-balloon Enteroscopy for Obscure Small-bowel Bleeding
Acronym: DBE;SBE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Jian Shi, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ERK-2
Record Dates: First submitted 2010-07-28; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-07

CONDITIONS: Small-Bowel Disorders
Keywords: Small-Bowel Disorders; Double-balloon enteroscopy; Single-balloon enteroscopy
MeSH Terms: interventions — Double-Balloon Enteroscopy; Single-Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double-balloon enteroscopy (Active Comparator): DBE for suspected or known small-bowel bleeding
  Interventions: Procedure: Double-balloon enteroscopy
- Single-balloon enteroscopy (Active Comparator): SBE for suspected or known small-bowel bleeding
  Interventions: Procedure: Single-balloon enteroscopy

INTERVENTIONS:
Procedure: Double-balloon enteroscopy — Double-balloon enteroscopy
  Arms: Double-balloon enteroscopy
Procedure: Single-balloon enteroscopy — Single-balloon enteroscopy
  Arms: Single-balloon enteroscopy

SUMMARY:
Double-balloon enteroscopy (DBE) is now an established method for diagnostic and therapeutic small-bowel endoscopy. Single-balloon enteroscopy (SBE) has been introduced to simplify the technique. A prospective randomized study was carried out to compare the two methods in obscure small bowel bleeding

DETAILED DESCRIPTION:
Th e double-balloon enteroscopy (DBE) system, developed by Dr Yamamoto, was presented for the fi rst time in Japan in 2001. The system has become established throughout the world for diagnostic and therapeutic small-bowel examinations, and it is now used universally in routine clinical work.

Another balloon enteroscopy system was recently introduced in which only one balloon is attached at the tip of the overtube; the method is therefore known as SBE. SBE is a simplification of the double balloon method, and its value has already been confirmed for difficult colonoscopies. The question of whether similar results can be achieved with the single balloon method in the more complex situation of the small bowel has not yet been answered.

ELIGIBILITY:
Inclusion Criteria:

1. suspected or known small-bowel bleeding
2. age: 16-70

Exclusion Criteria:

1. pregnancy
2. coagulation disorders
3. prior surgery of the small bowel and colon

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
whether the complete enteroscopy is achieved? | 2 hours
  the rate of complete enteroscopy in both groups.

SECONDARY OUTCOMES:
Preparation time | 2 hours
Investigation time | 2 hours
side effects | 2 days
Diagnostic yield | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jian Shi, MD, Principal Investigator — Shanghai Changzheng Hospital; Bin Shi, MD, Principal Investigator — Shanghai Changzheng Hospital; Wei-Fen Xie, MD, Study Director — Shanghai Changzheng Hospital
Locations (1):
- Shanghai changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Frantz DJ, Dellon ES, Grimm IS, Morgan DR. Single-balloon enteroscopy: results from an initial experience at a U.S. tertiary-care center. Gastrointest Endosc. 2010 Aug;72(2):422-6. doi: 10.1016/j.gie.2010.03.1117. Epub 2010 Jun 11. PMID 20541189
- [Result] May A, Farber M, Aschmoneit I, Pohl J, Manner H, Lotterer E, Moschler O, Kunz J, Gossner L, Monkemuller K, Ell C. Prospective multicenter trial comparing push-and-pull enteroscopy with the single- and double-balloon techniques in patients with small-bowel disorders. Am J Gastroenterol. 2010 Mar;105(3):575-81. doi: 10.1038/ajg.2009.712. Epub 2010 Jan 5. PMID 20051942